CLINICAL TRIAL: NCT00175669
Title: Randomized Controlled Trial of a Botulinum A Toxin (Botox) Injection in the Gastrocnemius Muscle in Children With Idiopathic Toe Walking
Brief Title: Trial of a Botulinum A Toxin (Botox) Injection in the Gastrocnemius Muscle in Children With Idiopathic Toe Walking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Christine Alvarez, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C00-0160; CW: 00-0500
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Idiopathic Toe Walking
Keywords: Randomized control trial; placebo-control study

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botox injections — Data not known.

SUMMARY:
The purpose of this study is to compare the effect of Botox and casting to placebo and casting for reducing toe walking problems in children who are idiopathic toe walkers.

DETAILED DESCRIPTION:
Patients who have been seen by one of the 5 paediatric orthopaedic surgeons at British Columbia's Children's Hospital and have been referred to the Shriner's gait lab for assessment of idiopathic toe walking will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been seen by one of the 5 paediatric orthopaedic surgeons at British Columbia's Children's Hospital and have been referred to the Shriner's gait lab for assessment of idiopathic toe walking
* Clinical toe walkers - toe walkers as per gait lab's definition (loss of 1st ankle rocker, early heel rise [prior to 30% of the cycle] and A1 kinematic data)
* Aged 5 - 15 years old
* Parents and patients educated about protocol and willing to partake
* Cooperative patient with gait analysis and injection

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be based on gait analysis data - specifically whether post injection gait analyses show a reduction in the features that were used to determine the severity of the subjects' toe walking problem. | Data not known

SECONDARY OUTCOMES:
Ankle range of motion (dorsiflexion and plantarflexion) | collected at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada